CLINICAL TRIAL: NCT03581994
Title: Drug-Drug Interaction (DDI™) Effectiveness and Clinical Awareness Randomized Controlled Trial
Brief Title: DDI Effectiveness and Clinical Awareness
Acronym: DECART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Aegis Sciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00024720
Record Dates: First submitted 2018-06-18; First posted 2018-07-10 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Drug-Drug Interactions

STUDY DESIGN:
Intervention Model Description: Two-arm parallel intervention assignment using identical educational materials but different question prompt approaches. Control arm included.
Who Masked: Care Provider
Masking Description: Single-blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Practice (No Intervention): Not receiving any intervention/educational materials on drug-drug interaction testing
- Compulsory DDI Testing (Experimental): Receiving educational materials on drug-drug interaction testing and a sample test report when caring for patient cases.
  Interventions: Diagnostic Test: DDI Test Report
- Optional DDI Testing (Experimental): Receiving educational materials on drug-drug interaction testing and given a sample test report if ordered when caring for patient cases.
  Interventions: Diagnostic Test: DDI Test Report

INTERVENTIONS:
Diagnostic Test: DDI Test Report — Test results of simulated patients
  Arms: Compulsory DDI Testing; Optional DDI Testing

SUMMARY:
The DECART study will determine if primary care physicians, including internists and family physicians, are able to identify and address drug-drug interactions among simulated patients and whether those physicians, when given access to Aegis Drug-Drug Interaction test results, improve patient management, take steps to reduce DDI risk, and optimize unnecessary resource utilization.

DETAILED DESCRIPTION:
The DECART study is a pre-post, two round, randomized controlled study of a nationally representative sample of 330 primary care physicians randomly assigned to a control or one of two intervention arms. Once eligibility is determined and providers are enrolled in the study, they will be asked to complete a questionnaire describing their practice and professional background. They will then care for a total of 6 CPV® simulated patients. The simulated patients will be adults aged 30-75 and present with various clinical conditions and potential drug interactions. The design and intervention consists of two rounds with an intervention among two thirds of the participants.

* Round 1 (Baseline Assessment): Providers in both the control and intervention groups will care for 3 CPV simulated patients using their standard practice approach, to evaluate their awareness of DDI interactions and associated variability in caring for patients at risk for DDIs.
* Intervention/DD! Education: Approximately 3 weeks after CPV Round 1 is complete, the intervention arms will receive Aegis test education materials, consisting of: 1) on-demand, online video on the Aegis DDI test, 2) example test results, 3) example case study, 4) clinical care reference guide, and 5) test overview.
* Round 2 (Post-Educational Intervention Assessment): Approximately 3 weeks after the intervention, all providers in the control and intervention arms will receive another 3 simulated patients to care for to determine if their awareness has changed and if their practice has improved. In the post--educational assessment, one-half of intervention participants will have access to Aegis DDI test results for their patients to help guide their decision making. The other half will have the option of receiving test results if ordered. Control physicians will continue to their standard practice approach.

ELIGIBILITY:
Inclusion Criteria:

1. Provide consent to participate in the study
2. Board-certified physician currently practicing in the following areas:
3. Internal medicine
4. Family medicine
5. Have practiced as a board-certified physician in internal or family medicine for greater than 2 but less than 30 years.
6. Have not used Aegis DDI
7. English-speaking
8. Community/ non-academic based practice setting
9. 40 patients under care weekly
10. 15% of their patient panel on opioid pain medications
11. Access to the internet

Exclusion Criteria:

1. Provide consent to participate in the study
2. Board-certified physician currently practicing in the following areas:
3. Internal medicine
4. Family medicine
5. Have practiced as a board-certified physician in internal or family medicine for greater than 2 but less than 30 years.
6. Have not used Aegis DDI
7. English-speaking
8. Community/ non-academic based practice setting
9. 40 patients under care weekly
10. 15% of their patient panel on opioid pain medications
11. Access to the internet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Drug-Drug Interaction (DDI) diagnosis | 3 months
  Difference in difference between the control and the intervention group in their identification and effective treatment of DDls.

SECONDARY OUTCOMES:
Quality of care | 3 months
  Difference in difference between the control and the intervention groups in the overall quality of care as measured by their combined domain and individual item CPV scores (ranging from 0% to 100%) for the 9 patient types in aggregate and by case type.
DDI adoption | 3 months
  Rate of DDI adoption after receiving educational material on the benefits of testing in patients who are at risk.
Resource utilization | 3 months
  Difference in health care utilization and/or costs in patients tested with DDI versus the control group in aggregate and by case type.

CONTACTS AND LOCATIONS:
Overall Officials: John W Peabody, MD PhD, Principal Investigator — President
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared